CLINICAL TRIAL: NCT03298919
Title: Efficacy of Exercise Videogames for Physical Activity Adoption and Maintenance
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Miriam Hospital (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 203711; R01HL109116 (NIH)
Record Dates: First submitted 2017-09-27; First posted 2017-10-02 (Actual); Last update posted 2019-04-25 (Actual); Status verified 2017-09

CONDITIONS: Physical Activity
MeSH Terms: conditions — Motor Activity | interventions — Exercise

STUDY DESIGN:
Intervention Model Description: 3-group design
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Exercise Videogames (Experimental): Exercise videogames 3 times weekly for 12 weeks followed by 6 months of home practice
  Interventions: Behavioral: Exercise Video Games; Behavioral: Home exercise videogames
- Standard Exercise (Active Comparator): Exercise using aerobic equipment such as stationary bikes and treadmills 3 times weekly for 12 weeks followed by home practice
  Interventions: Behavioral: Aerobic Exercise; Behavioral: Home Standard Exercise
- Wellness Control (No Intervention): Weekly mailings on general health and wellness topics for 12 weeks followed by monthly mailings for 6 months.

INTERVENTIONS:
Behavioral: Exercise Video Games — 12 weeks laboratory based exercise videogames
  Arms: Exercise Videogames
Behavioral: Aerobic Exercise — Stationary bike and/or treadmill walking for 12 weeks
  Arms: Standard Exercise
Behavioral: Home exercise videogames — videogame console and active videogames
  Arms: Exercise Videogames
Behavioral: Home Standard Exercise — Personalized physical activity promotion materials
  Arms: Standard Exercise

SUMMARY:
This is a 3-arm trial to compare exercise videogames versus traditional standard exercise using stationary bikes and treadmills versus a control condition. Results will examine minutes of physical activity at 12 weeks and 6 month follow up between conditions. We will also examine changes in indicators of cardiovascular health (e.g., body mass index, lipids) and changes in psychological factors that may be predictive of continued exercise engagement.

DETAILED DESCRIPTION:
To test the efficacy of a 12-week supervised, laboratory based program of an exercise videogame (EVG) program to increase time spent in moderate-to-vigorous physical activity (MVPA) and improve cardiovascular health and fitness indices compared to Standard and Control programs. Participants will be randomly assigned to (1) a supervised program of Exercise Videogames (EVG); (2) a supervised standard exercise program (Standard), using aerobic exercise equipment (e.g., treadmill, stationary bike); or (3) a Control condition. We will also examine the effect of home-based exercise videogames compared to a home-based standard PA program on MVPA maintenance during the 6-month follow up period. We will examine changes in cardiorespiratory fitness (i.e., estimated VO2max), blood pressure, resting heart rate, body composition and blood lipids at baseline, week 12 and at 6-months follow up. We will also examine changes in theoretically-based cognitive and affective constructs associated with physical activity including: enjoyment, outcome expectations, self-efficacy, motivation, and goal-orientation.

ELIGIBILITY:
Inclusion Criteria:

* age > 18,
* In generally good health
* No medical conditions that would interfere with exercise
* Currently engaging in less than 60 minutes of physical activity per week

Exclusion Criteria:

* body mass index over 40
* current or planned pregnancy
* hospitalization from a physical or mental disorder in the past 6 months
* hypertension (defined as: blood pressure ≥ 140/90)
* anti-hypertensive medication
* medications that may impair physical activity tolerance (e.g., beta blockers)
* current cardiovascular disease
* current pulmonary disease
* diabetes
* thyroid disorders
* renal or liver disease
* orthopedic conditions that would prevent or limit exercise

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 283 (Actual)
Dates: Start 2012-09-01 (Actual); Primary Completion 2016-08-29 (Actual); Study Completion 2017-09-30 (Actual)

PRIMARY OUTCOMES:
MVPA | 12 weeks
  moderate to vigorous physical activity minutes
MVPA Maintenance | 6 months
  moderate to vigorous physical activity minutes

CONTACTS AND LOCATIONS:
Overall Officials: Beth Bock, PhD, Principal Investigator — The Miriam Hospital
Locations (1):
- The Miriam Hospital- CORO building, Providence, Rhode Island, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Serber ER, Ciccolo J, Palmer K, Cobb V, Tilkemeier PL, Bock BC. The feasibility of exercise videogames for cardiovascular risk reduction among adults: a pilot for "Wii heart fitness". J Sports Med Phys Fitness. 2016 Mar;56(3):319-27. Epub 2015 Feb 18. PMID 25692860
- [Result] Bock BC, Thind H, Dunsiger SI, Serber ER, Ciccolo JT, Cobb V, Palmer K, Abernathy S, Marcus BH. Exercise videogames for physical activity and fitness: Design and rationale of the Wii Heart Fitness trial. Contemp Clin Trials. 2015 May;42:204-12. doi: 10.1016/j.cct.2015.04.007. Epub 2015 Apr 17. PMID 25896114
- [Result] Bock BC, Dunsiger SI, Ciccolo JT, Serber ER, Wu WC, Tilkemeier P, Walaska KA, Marcus BH. Exercise Videogames, Physical Activity, and Health: Wii Heart Fitness: A Randomized Clinical Trial. Am J Prev Med. 2019 Apr;56(4):501-511. doi: 10.1016/j.amepre.2018.11.026. Epub 2019 Feb 16. PMID 30777705
- [Derived] Bock BC, Dunsiger SI, Ciccolo JT, Serber ER, Wu WC, Sillice M, Marcus BH. Mediators of physical activity between standard exercise and exercise video games. Health Psychol. 2019 Dec;38(12):1107-1115. doi: 10.1037/hea0000791. Epub 2019 Sep 12. PMID 31512923